CLINICAL TRIAL: NCT07140380
Title: Phase 2b, Proof-of-Concept, Single-center, Double-Masked, Randomized Study Comparing the Safety, Tolerability, and Efficacy of Three Different Ophthalmic Eyelid Wipe Dosing Techniques Using IVW-1001 in Subjects With Dry Eye Disease
Brief Title: Phase 2b Controlled Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IVIEW Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IVW-1001-CS-202
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye Disease
Keywords: dry eye disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Randomized cross-over to one of three dosing techniques with interperiod washout of 14 days.
Who Masked: Outcomes Assessor
Masking Description: All site personnel will be aware of the assigned IVW-1001 Ophthalmic Eyelid Wipe 0.2% concentration. However, subjects will be randomized to the sequence of the assigned dosing technique procedures which will be provided to individual subjects by the unmasked dosing technique coordinator only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- IVW-1001 Ophthalmic Wipe - Method 1 (Experimental): With eyes completely closed, the subject should wipe upper eyelid in a nasal to temporal direction with the IVW-1001 Ophthalmic Eyelid Wipe while applying moderate pressure to the eyelid skin slightly away from the eyelash line.
  Interventions: Drug: IVW-1001 Ophthalmic Eyelid Wipe
- IVW-1001 Ophthalmic Wipe - Method 2 (Experimental): With eyes completely closed, the subject should wipe the upper eyelid in a nasal to temporal direction with the IVW-1001 Ophthalmic Eyelid Wipe while applying moderate pressure directly at the lash margin covering the eyelash line.
  Interventions: Drug: IVW-1001 Ophthalmic Eyelid Wipe
- IVW-1001 Ophthalmic Wipe - Method 3 (Experimental): With eyes completely closed, the subject should lay the IVW-1001 Ophthalmic Eyelid Wipe on the upper eyelid for 5 seconds, especially over the lash margin covering the eyelash line, then wiping the upper eyelid in a nasal to temporal direction. while applying moderate pressure directly at the lash margin covering the eyelash line .
  Interventions: Drug: IVW-1001 Ophthalmic Eyelid Wipe

INTERVENTIONS:
Drug: IVW-1001 Ophthalmic Eyelid Wipe — Dry eye treatment

SUMMARY:
Double-masked two period controlled trial of three eyelid wipe dosing techniques

DETAILED DESCRIPTION:
This is a randomized, single center, single -masked study to evaluate the safety, tolerability, and efficacy of IVW-1001 Ophthalmic Eyelid Wipe dosing techniques in subjects with DED. Treatments will be IVW 1001 Ophthalmic Eyelid Wipe 0.2% (low dose) and 0.4% (high dose). Subjects will participate in a 50-day, double -masked three dosing technique comparisons period using IVW-1001 Ophthalmic Eyelid Wipe 0.2% followed by a 14-day between period washout.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported diagnosis of DED in one or both eyes
* BCVA +0.70 logarithm of minimum angle of refraction (Snellen equivalent 20/100) or better in each eye at the Screening Visit
* For women of childbearing potential, confirmed negative pregnancy test at the Screening Visit, not nursing a child, and willing to comply with one of the acceptable methods of birth control described in the protocol
* History (by subject recollection) of artificial tear use within 30 days prior to the Screening Visit
* Unanesthetized Schirmer's test score 5-19 mm inclusive in at least 1 eye (same eye) at the Screening Visit and the Baseline Visit

Exclusion Criteria:

* Corneal fluorescein staining score of 4 in either eye in any zone using the National Eye Institute grading system at either the Screening Visit or the Baseline Visit
* IOP ≥23 mmHg in either eye at either the Screening Visit or the Baseline Visit
* History of glaucoma or ocular hypertension in either eye requiring past or current medical or surgical intervention

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tear production | Day 8 for each treatment
  Mean change from baseline in Unanesthetized Schirmer score

SECONDARY OUTCOMES:
Visual acuity | Day 8 for each treatment
  Mean change from baseline in Best Corrected Visual Acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Research Foundation, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No